CLINICAL TRIAL: NCT04745078
Title: Evaluation of the Use of Carboxytherapy in Periorbital Dark Circles
Brief Title: Carboxytherapy for Periorbital Dark Circles
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Principal Investigator, Heba Mahmoud, principal investigator, Alexandria University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0104074
Record Dates: First submitted 2021-02-03; First posted 2021-02-09 (Actual); Last update posted 2021-11-04 (Actual); Status verified 2021-11

CONDITIONS: Periorbital Disorder
Keywords: carboxytherapy; dark circles

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Carboxy30 (Active Comparator): carboxy30
  Interventions: Other: Caboxy30
- Carboxy60 (Active Comparator): carboxy60
  Interventions: Other: Caboxy60

INTERVENTIONS:
Other: Caboxy30 — carboxy30 to periorbital dark halos
  Other Names: Carboxy30
  Arms: Carboxy30
Other: Caboxy60 — carboxy60 to periorbital dark halos
  Arms: Carboxy60

SUMMARY:
the study evaluates carboxytherapy for the treatment of periorbital dark circles

DETAILED DESCRIPTION:
two different concentrations of carboxytherapy administered to patients are compared regarding efficacy

ELIGIBILITY:
Inclusion Criteria:

* healthy individuals with dark circles

Exclusion Criteria:

* infections, scarring, pregnancy, allergy, on treatment for the condition.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2021-04-01 (Actual); Study Completion 2021-05-15 (Actual)

PRIMARY OUTCOMES:
Improvement of Melanin index | 6 weeks
  change in melanin index of the dark circles
Improvement of erythema index | 6 weeks
  change in erythema index of the dark circles

CONTACTS AND LOCATIONS:
Overall Officials: Ossama H Roushdy, MD, Study Chair — University of Alexandria
Locations (1):
- Faculty of Medicine,Alexandria University, Alexandria, Egypt